CLINICAL TRIAL: NCT04907500
Title: Prospective Evaluation of the Clinical Safety and Effectiveness of Hydrophilic Acrylic Intraocular Lens
Brief Title: Prospective Evaluation of an Hydrophilic Acrylic Intraocular Lens
Acronym: UVEA 809
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LISA 809 BER-401-20
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cataract Senile
MeSH Terms: interventions — Lenses, Intraocular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multifocal IOL (Experimental): Implantation of a multifocal intraocular lens
  Interventions: Device: Intraocular lens

INTERVENTIONS:
Device: Intraocular lens — Cataract surgery

SUMMARY:
Evaluation of the clinical safety and effectiveness of an hydrophilic acrylic intraocular lens

DETAILED DESCRIPTION:
To show safety and the effectiveness in regard to the monocular corrected distance visual acuity (CDVA) and the distance-corrected near visual acuity (DCNVA) at 6 months postoperative.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of any gender, aged 18 years or older
2. Patient is planned for aged-related cataract surgery and implantation of the study IOL into the capsular bag in at least one eye
3. Patient is willing and capable of providing informed consent
4. Patient is willing and capable of complying with visits and procedures as defined by this protocol

Exclusion Criteria:

1. Preoperative corrected distance visual acuity (CDVA) better than 0.3 logMAR (0.5 decimal)
2. Endothelial cell count of less than 2000/mm2
3. Ocular disorder that could potentially cause a clinically significant future visual acuity loss
4. Preoperative corneal astigmatism ative corneal to be < 1 D.
5. Clinically significant anterior segment pathology (e.g. chronic uveitis, iritis, aniridia, rubeosis iridis, anterior membrane dystrophies, poor pupil dilation, etc.)
6. Clinically significant abnormal corneal finding (e.g. keratoconus, pellucid marginal degeneration, or irregular astigmatism, clinically significant corneal membrane dystrophies)
7. Any clinically significant condition that could affect IOL stability (e.g. zonular dialysis, evident zonular weakness or dehiscence, etc.)
8. Any History of clinically significant retinal pathologies or ocular diagnosis (e.g. diabetic retinopathy, ischemic diseases, macular degeneration, retinal detachment, optic neuropathy optic nerve atrophy, amblyopia, strabismus, microphthalmos, aniridia, epiretinal membrane etc.) that could alter or limit final postoperative visual prognosis
9. Any acute infection (acute ocular disease, external/internal infection, systemic infection)
10. Any previous intraocular and corneal surgery
11. Uncontrolled glaucoma or IOP higher than 24mmHg under ocular hypertension treatment
12. Current systemic or ocular pharmacotherapy that effects patients'vision
13. Current pathology or condition that could be a risk for the patient according to the investigator opinion
14. Women during pregnancy and/or lactation
15. Patients unable to meet the limitations of the protocol or likely of noncooperation during the trial
16. Patients whose freedom is impaired by administrative or legal order
17. Subject is enrolled in any other concurrent clinical study, with the exception of local mandatory governmental registries and observational studies/registries, that do not affect patients'vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-08-06 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Monocular corrected distance visual acuity (CDVA) | 6 months after the implantation
  Monocular corrected distance visual acuity measured in logMAR

CONTACTS AND LOCATIONS:
Locations (1):
- DUO STIL SRL , Clinica Oftalmologica Medoptic, Suceava, Romania